CLINICAL TRIAL: NCT03683316
Title: The Impact of Kangaroo Mother Care on Work of Breathing Indices and Oxygen Saturation Stability in Very Low Birth Weight Infants
Brief Title: Work of Breathing and Kangaroo Mother Care
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: DDD603995
Record Dates: First submitted 2018-05-08; First posted 2018-09-25 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Premature Infant; Work of Breathing; Oxygen Saturation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all infants: There will be one arm for this study. All infants will receive a similar intervention during their routine kangaroo mother care (KMC). KMC is a national and international standard of care. This is an observational study of how infants breath while participating in KMC compared to how they breath while in a crib or incubator. Work of breathing will be measured at baseline and then during KMC. Mothers will participate in KMC regardless of participation in the study. Work of breathing will be measured by using Respiratory Inductance Plethysmography (RIP). This scientifically measures work of breathing (specifically phase angles) by placing soft bands around the abdomen and chest. The actual "intervention" is a standard of care and something that the mother infant dyad will do regardless of the study. Each mother / infants pair is expected to be actively enrolled for approximately 2 hours.

SUMMARY:
To compare work of breathing and oxygen saturation before, during, and after kangaroo mother care in preterm very low birth weight (VLBW) infants stable on non-invasive respiratory support.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants (those less than 1500g at birth)
* Respiratory insufficiency
* >4d PMA
* Stable and receiving non-invasive respiratory support for ≥12 hours (NC, HFNC or CPAP)
* Requiring ≤40% supplemental FiO2

Exclusion Criteria:

* Infants with skeletal, neuromuscular or abdominal surgical disorders that may affect the accuracy of work of breathing measurements
* Infants who do not meet criteria to participate in kangaroo mother care

Ages: 4 Days to 6 Months | Sex: All
Age Groups: Child
Study Population: Very low birth weight infants in the NICU who meet inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change in work of breathing | 2 hours
  Work of breathing will be measured before, during, and after KMC. Comparisons will be made.

SECONDARY OUTCOMES:
Oxygen saturation | 2 hours
  Oxygen saturations will be measured before, during, and after KMC. Comparisons will be made.

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Kovatis, MD, Study Director — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Inc, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided